CLINICAL TRIAL: NCT03866356
Title: The Effectiveness of a Care Protocol Developed Using the Star Model on Female Patients With Stress Incontinence: A Randomized Controlled Trial
Brief Title: The Effectiveness of a Stress Incontinence Care Protocol
Acronym: SICP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Emel Gülnar, Research Assistant, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KU
Record Dates: First submitted 2019-03-02; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Stress Incontinence, Female; Nursing
Keywords: Nursing; evidence-based practice; Star model; stress incontinence; nursing care protocol; female
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group received care according to the SICP (Table 2). One of the researchers gave each participant one-on-one education in line with SICP. They were also provided with the booklet that had been prepared in accordance with SICP. The participants were phoned every week for eight weeks and offered counseling within the scope of SICP and then were reevaluated at the end of eight weeks (Post-intervention). The participants were followed from the eighth to the twelfth week without any intervention (4-week post-intervention).
  Interventions: Behavioral: intervention group
- Control group (No Intervention): The control group received no intervention during the eight-week intervention period. The control group received standard care. The women were given no educational materials.

INTERVENTIONS:
Behavioral: intervention group — The women in the intervention group were provided care according to SICP
  Arms: Intervention group

SUMMARY:
This study seeks to contribute to nursing practices by developing and stress incontinence care protocol with the help of the Star model and implementing this care protocol for the purpose of standardizing patient care outcomes.

DETAILED DESCRIPTION:
To identify the effectiveness of a care protocol developed using the Star model on outcomes in female patients with stress incontinence.

Information and evidence needs to be translated into nursing practice and applied to clinical decision-making in stress incontinence cases. Evidence-based study models such as the Star model provide guidance on using evidence to develop clinical guidelines and care protocols. The Star model is designed to improve patient outcomes by creating a bridge between research and clinical practice. There is currently no published stress incontinence care protocol based on the Star model. Although there is one published study of a care protocol for urinary incontinence, this protocol was not drawn up on the basis of an evidence-based model.

Women that matched the sample criteria were recruited into the study. After their consent was obtained, the women were randomized into an intervention and a control group. The women in the intervention group were provided care according to stress incontinence care protocol. The control group received no intervention during the eight-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were being female, ≥ 18 years, having an initial diagnosis of SI, being literate, having no sensory disorder affecting communication, and agreeing to participate in the research

Exclusion Criteria:

* The exclusion criteria were pregnancy, presence of a urinary tract infection and previous treatment for SI. The removal criteria were patient non-compliance with the protocol, failure in contacting the patient and the patient's wish to withdraw from the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
King's Health Questionnaire | 20 minutes
  This 32-item tool measures quality of life. Scores range from 0 - 100, with low scores indicating good quality of life.
Broome Pelvic Muscle Exercise Self-Efficacy Scale | 15 minutes
  This instrument was developed to measure perceived self-efficacy in pelvic floor muscle exercise. It consists of 23 items organized in two subscales. The total score ranges from 0 - 100 and scores are classified as follows: ≤ 32(low self-efficacy); 33 55 points (medium self-efficacy); ≥ 56 points (high self-efficacy).
Three-day voiding diary | 3 days
  This is a semi-objective tool used to record voiding frequency, amount of urine, amount and type of liquid intake, incontinence frequency and the frequency of pad-changing.
One-hour pad test | 1 hour
  This test provides an objective measure of the quantity of urine leakage in a one-hour period. Before the test, the dry pad is weighed using precision scales and this weight is deducted from the wet weight to give the weight of leaked urine (Krhut et al., 2014). First the patient is given the pre-weighed pad and is then asked to drink 500 cc water and to rest in a seated position for a half-hour. In the following half- hour, the patient stands up and sits down 10 times, coughs 10 times, runs in place for 1 minute, bends to pick something up from the floor 5 times, and then climbs a flight of stairs. After one hour, the pad is taken from the patient and re-weighed on the same precision scales. The weight of the dry pad is deducted from the weight of the wet pad and the weight of urine is recorded.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kaya S, Akbayrak T, Toprak Celenay S, Dolgun A, Ekici G, Beksac S. Reliability and validity of the Turkish King's Health Questionnaire in women with urinary incontinence. Int Urogynecol J. 2015 Dec;26(12):1853-9. doi: 10.1007/s00192-015-2786-6. Epub 2015 Jul 26. PMID 26209953
- [Background] Krhut J, Zachoval R, Smith PP, Rosier PF, Valansky L, Martan A, Zvara P. Pad weight testing in the evaluation of urinary incontinence. Neurourol Urodyn. 2014 Jun;33(5):507-10. doi: 10.1002/nau.22436. Epub 2013 Jun 24. PMID 23797972
- [Background] Stevens KR. The impact of evidence-based practice in nursing and the next big ideas. Online J Issues Nurs. 2013 May 31;18(2):4. PMID 23758422
- [Background] Schaffer MA, Sandau KE, Diedrick L. Evidence-based practice models for organizational change: overview and practical applications. J Adv Nurs. 2013 May;69(5):1197-209. doi: 10.1111/j.1365-2648.2012.06122.x. Epub 2012 Aug 9. PMID 22882410
- [Background] Zengin N, Pinar R. Reliability and validity of the continence self-efficacy scale in Turkish women with urinary incontinence. Nurs Health Sci. 2012 Sep;14(3):277-84. doi: 10.1111/j.1442-2018.2012.00692.x. Epub 2012 May 27. PMID 22632069